CLINICAL TRIAL: NCT03925519
Title: Supervised Aerobic Exercise as Anti-adiposity and Cardioprotective Modulates in Patients With Type 2 Diabetes Mellitus
Brief Title: Exercise as Cardio Protective Modulates in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sami Gabr, clinical Professor, King Saud University
Other Study IDs: RRC-2013-010
Record Dates: First submitted 2019-04-17; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus; Exercise
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples were obtained from all subjects at 0800 h after an overnight fast before and after the training program Venous blood samples (5 mL) were collected into plain tubes, the samples were allowed to clot for half an hour following which samples were centrifuged for 15 minutes at 2000 rpm. Samples were given a coded study identification number and were stored frozen at 80°C until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-obese: non-obese diabetic patients (n= 25, BMI ≤ 30 kg/m2) were subjected to supervised aerobic exercise
- obese group: obese diabetic group (n= 25, BMI ≥ 30 kg/m2)
  Interventions: Other: Supervised aerobic exercise

INTERVENTIONS:
Other: Supervised aerobic exercise
  Groups: obese group

SUMMARY:
* Physical exercise for 6 months produced significant improvement in adiponectin, hs-CRP, and nitric oxide (NO) and was significantly correlated with adiposity markers, lipid profile and glycemic control factors in both obese and non-obese diabetic patients.
* Patients with good physical activity reported a significant decrease in BMI, CHD risk scores, reduced hs-CRP, an increase in the levels of adiponectin and nitric oxide.
* In patients with type 2 diabetes mellitus, adiposity markers, lipid profile, hs-CRP, and adiponectin were significantly improved following moderate exercise interventions

DETAILED DESCRIPTION:
To elucidate the potential role of exercise as anti-adiposity and anti-cardio protective modulates, we thought to investigate the effect of supervised aerobic training of moderate intensity on adiposity markers, nitric oxide level, plasma adiponectin, hs-CRP, and its association with CHD risk score in obese and non-obese patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes for more than 5 years.
* Patients who were diagnosed according to the criteria of the American diabetes association.
* Not receiving any drugs affecting the data obtained
* had Normal daily diets
* Not participating in any other exercise programs
* Without any musculoskeletal disorders affecting an exercise program

Exclusion Criteria:

* Exclusion criteria included anemia, overt complications of diabetes like nephropathy, neuropathy, retinopathy, obvious ischemic heart disease (angina, myocardial infarction, and lead electrocardiogram abnormalities), HCV, HBV, chronic liver and kidney diseases, hypothyroidism, and drugs (diuretics; oral contraceptives).

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty subjects diagnosed with type 2 diabetes for more than 5 years aged 45-70 years were invited in the period from 2013 to 2014 to participate in this study. Patients were diagnosed according to the criteria of American diabetes association.32 Based on the values of BMI, the patients were classified into two groups, obese diabetic group (n= 25, BMI ≥ 30 kg/m2) and non-obese group (n= 25, BMI ≤ 30 kg/m2).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-01-25 (Actual); Primary Completion 2014-04-15 (Actual); Study Completion 2014-05-26 (Actual)

PRIMARY OUTCOMES:
Estimation of coronary heart disease risk score | six months
  The incidence risk score of coronary heart disease among type 2 diabetic participants .patients were classified into T2DM patients with high CHD risk (UKPDS risk ; ≥ 20%), moderate CHD risk (UKPDS risk ; 10-20%), and low (UKPDS risk;< 10%) .
Analysis of blood sugar, glycated hemoglobin (HbA1c) | six months
  Blood glucose was measured using a glucose oxidase and peroxidase (GOD-POD) colorimetric method before and after exercise training

SECONDARY OUTCOMES:
Analysis of Nitric Oxide | six months
  Plasma NO concentration was estimated as nitrate and nitrite using High Performance Liquid Chromatography technology (HPLC). Patients were subjected for nitri oxide analysis before and after exercise training interventions